CLINICAL TRIAL: NCT00437398
Title: Islet Transplantation for Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to difficulty in recruiting subjects, and ran short of funds.
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Yogish C. Kudva, MBBS, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-003564; UL1RR024150 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: hypoglycemic unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Transplant (Experimental): Subjects will receive standard intraportal transplantation or portal venous system infusion via laparotomy of purified pancreatic islets.
  Interventions: Biological: Islet Transplant

INTERVENTIONS:
Biological: Islet Transplant — Purified pancreatic islets

SUMMARY:
The complex program of insulin replacement for type 1 diabetes that is current clinical standard of care is difficult to implement for long periods of time, associated with an increased risk of severe hypoglycemia and implemented by less than 50 % of the population of such patients. Outcomes of transplantation of isolated human islets have substantially improved and been performed at about 40 institutions around the world. We are proposing a clinical phase 1/phase 2 study of islet transplantation alone evaluating safety and efficacy in five patients with type 1 diabetes. Islet isolation from deceased donor pancreases will be performed at the Mayo Rochester Islet Isolation facility and islets infused by Interventional Radiology into the portal venous system. Following islet infusion, patients will be hospitalized for 48 hours in the General Clinical Research Center (GCRC) or at the Rochester Methodist Hospital. Multiple safety and efficacy outcomes will be followed on multiple occasions during the first year and periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Duration of diabetes: 5 years or more
* Type 1 diabetes with C-peptide < 200 pmol/L and a simultaneous plasma glucose between 60 and 250 mg/dl
* Complex insulin program supervised by an endocrinologist for at least 6 months
* Hypoglycemic unawareness diagnosed using Clarke Awareness Questionnaire
* Body weight < 70 kg
* Body Mass Index < 30 kg/m^2
* Insulin requirement < 40 units/day by multiple daily injections or < 30 units /day by external insulin pump or < 0.6 unit/kg/day with a HbA1c < 7.0 % ( Normal < 6 %)
* No overt cardiovascular disease
* No laser treatment for retinopathy
* Retinopathy diagnosed by ophthalmologist to be stable and requiring no further evaluation for at least one year
* Women of child bearing age will have a negative pregnancy test at screening and time of trial initiation
* Women enrolled in the trial should be willing to practice birth control while on immunosuppression
* No psychologic issues that would interfere with adherence to safe clinical practice
* Blood type (ABO) compatibility
* No evidence of chronic liver disease (aspartate aminotransferase (AST) < 2.5 times normal, alanine aminotransferase (ALT) < 2.5 times normal, international normalized ratio (INR) < 1.4, No evidence of fatty liver on abdominal ultrasound.

Exclusion Criteria:

* Ongoing infection
* Ongoing alcohol or drug abuse
* Clinical portal hypertension
* Gall stones
* Liver hemangioma on ultrasound interfering with islet infusion
* Lack of updated immunization
* Unstable cardiovascular status as defined by:

  1. Myocardial infarction/acute coronary syndrome in last year
  2. Significant coronary atherosclerosis on angiography
  3. Active ischemia at evaluation
* Pre-trial low-density lipoprotein (LDL) cholesterol > 100 and triglycerides > 200 mg/dl with or without lipid lowering therapy
* Active peptic ulcer disease
* Previous organ transplantation except islet transplantation
* Negative serology for Epstein-Barr Virus (EBV) or ongoing acute EBV infection
* Previous malignancy unless

  1. 5 years ago
  2. basal cell cancer
  3. squamous cell cancer
* Requiring steroid therapy for any reason
* Positive Purified Protein Derivative (PPD - Tuberculosis Skin Test)
* Serological evidence of HIV, Hepatitis C or Hepatitis B
* Chronic anemia
* Single Antigen B (SAB) normalized value >1500
* Renal disease

  1. Iothalamate clearance < 70 cc/min
  2. 24 hour urine protein > 500 mg/24 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogish C. Kudva, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: Three subjects were screened for islet transplantation; one subject was ineligible, being Epstein-Barr virus (EBV) seronegative.
Period: Overall Study
Arm/Group | Islet Transplant
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplant
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Hypoglycemic Events After Transplant
Description: Hypoglycemia is an abnormally diminished content of glucose in the blood.
Time Frame: 3, 6, 9, and 12 months since islet transplantation
Population: The sample size (n=2) was too small to perform a meaningful analysis; therefore the data were not analyzed due to study termination.
Arm/Group | Islet Transplant
Number analyzed (Participants) | 0

2. Secondary Outcome: Mean Glycated Hemoglobin (HbA1c) Since Transplant
Description: HbA1c is a lab test that shows the average level of blood sugar (glucose) over the previous 3 months. It shows how well the subject is controlling his/her diabetes.
Time Frame: 3, 6, 9, and 12 months since islet transplantation
Population: as for outcome 1
Arm/Group | Islet Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Subjects were hospitalized for 48 hours for the transplant. They stayed close to hospital for 10-14 days for followup. Subjects were clinically evaluated every 3 months for the first year and annually thereafter.
Arm/Group | Islet Transplant
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplant (N=2)
Hospitalization due to neutropenia and fever (Infections and infestations) | 1 (1) — Six months after transplant, subject 2 developed neutropenia and was admitted to the hospital for 2 days following a 3 day illness of fever, chills, nausea, emesis and body aches. The subject received 3 doses of neupogen.
hemodynamic instability (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplant (N=2)
Hypoglycemia (Endocrine disorders) | 1 (2)
Mild change in liver function tests (Injury, poisoning and procedural complications) | 1 (1) — Subject 1 experienced dental caries requiring extraction on day 40 after procedure 1. This required Cephalexin administration resulting in a mild change in liver function tests.

LIMITATIONS AND CAVEATS:
The study was terminated early due to difficulty in recruiting subjects, and ran short of funds. The sample size (n=2) was too small to perform a meaningful analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No